CLINICAL TRIAL: NCT02162394
Title: Study to Determine the Feasibility of Wireless Electrocardiography
Brief Title: A Study to Determine the Feasibility of Wireless Electrocardiography
Status: Completed | Type: Observational
Sponsor: Peerbridge Health, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-022A
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation; Premature Atrial and Ventricular Beats; Conduction Defects; Normal Sinus Rhythm
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Referred for Holter monitoring
  Interventions: Device: Observational ambulatory ECG monitoring

INTERVENTIONS:
Device: Observational ambulatory ECG monitoring

SUMMARY:
The investigators are conducting a prospective, observational study to examine the ECG waveforms captured by the new medical device as compared to a traditional Holter monitor for subsequent use in visual diagnoses of atrial and ventricular arrhythmias as well as cardiac impulse and/or conduction disorders by qualified clinicians.

The hypothesis is that this new medical device prototype is non-inferior to traditional Holter monitoring for capturing ECG waveforms that can be visually assessed for atrial and ventricular arrhythmias as well as disorders of cardiac impulse formation and/or conduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Patients must have a medical indication to wear a Holter monitor
* Patients must not be pregnant
* Patients must be able to comply with the study procedures
* Patients must be willing to participate and able to provide informed consent
* Patients must be willing to wear both devices (Holter and the wireless device prototype) simultaneously and continuously for a 2 to 3 hr period

Exclusion Criteria:

* Patients who are not able or willing to comply with study procedures
* Patients with an existing implanted cardioverter-defibrillator and/or pacemaker
* Patients with a known life threatening arrhythmia
* Patients who manifest low voltage on their electrocardiogram
* Patients affected by inflammatory and/or infectious skin disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred for 24 hour Holter monitoring
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percent of 8 second ECG strips of sufficient quality for visual diagnosis | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No